CLINICAL TRIAL: NCT01258881
Title: Retrospective Study of Ovarian Cancer Patients With Brain Metastasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Wen-Fang Cheng/Professor, National Taiwan University Hospital
Other Study IDs: 201004066R
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Last update posted 2010-12-13 (Estimated); Status verified 2010-12

CONDITIONS: Ovarian Cancer; Brain Metastases
MeSH Terms: conditions — Ovarian Neoplasms; Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Ovarian cancer, especially epithelial ovarian carcinoma, has the highest mortality rate among the gynecologic malignancies. The majority of patients with epithelial ovarian carcinoma are diagnosed at advanced stage which has the overall survival rates of only 19-30%. As the advance in the managements which prolonged the overall survival, metastatic lesion in rare location such as brain was noted in few patients of ovarian cancer in recent years. In the retrospective study, the investigators will review the medical records of the ovarian cancer patients with brain metastasis in the investigators hospital to investigate the incidence, clinical courses, optimal managements and possible prognostic factors in the rare condition.

DETAILED DESCRIPTION:
The ovarian cancer patient treated at the Department of Obstetrics and Gynecology of the National Taiwan University Hospital were retrospectively collected. The cancer registration database was searched for the patients with ovarian carcinoma who brain metastases were also diagnosed. The medical records of these patients were reviewed with particular attention to the results of histo-pathological and radiologic reports. Patients with other synchronous primary brain tumor were excluded. The initial management of primary tumor, including the surgery and adjuvant chemotherapy, and the clinical courses and disease status, such as remission, recurrence and progression, were all carefully reviewed. The intra-cranial lesions were all diagnosed by imaging studies, including brain computed tomography (CT) and magnetic resonance imaging (MRI) scans. Therapeutic strategies for the metastatic lesions in the brain were also reviewed. All statistical analyses were performed using the SPSS 13.0 statistical software for Windows. P<0.05 was defined as statistical significance. Survival was measured from the time of initial diagnosis of brain metastasis until the date of death or last contact, and was presented by Kaplan-Meier curves.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ovarian cancer and brain metastasis
* Patients ovarian cancer from National Taiwan University Hospital

Exclusion Criteria:

* none

Ages: 25 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ovarian cancer patients with brain metastasis
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Fang Cheng, Professor, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan